CLINICAL TRIAL: NCT02518958
Title: A Phase I, Open-Label, Multiple Ascending Dose Study to Assess the Safety and Tolerability of RRx-001 and Nivolumab in Subjects With Advanced Solid Tumors or Lymphomas For Which There Are No Currently Accepted Life-Prolonging Therapies (PRIMETIME)
Brief Title: A Phase I, Open-Label, Multiple Ascending Dose Study of RRx-001 and Nivolumab
Acronym: PRIMETIME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-14-02
Record Dates: First submitted 2015-08-04; First posted 2015-08-10 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Malignant Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — RRx-001; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RRx-001 + Nivolumab (Experimental): Patients enrolled in this trial will receive study drug (RRx-001) on Day 1 as a single agent. Nivolumab (3 mg/kg) will be administered on Day 2 or Day 3 as a single agent.
  Interventions: Drug: RRx-001; Drug: Nivolumab

INTERVENTIONS:
Drug: RRx-001
Drug: Nivolumab

SUMMARY:
This is a dose escalation protocol to determine the feasibility of co-administration of RRx-001 and nivolumab. Immune surveillance is an endogenous mechanism to cause remission of neoplastic growth. Epigenetic agents like RRx-001 are associated not only with enhanced gene transcription and restored expression of silenced genes but also with increased expression of pro-inflammatory mediators, upregulation of PD-L1 on tumor cells and de-repression of antigens that promote immune recognition of tumors. It is hypothesized that RRx-001, will prime or sensitize to immune checkpoint therapy targeting PD-1 interaction with nivolumab.

DETAILED DESCRIPTION:
This is an open-label dose escalation study, consisting of the following periods:

* 1) Screening Period (Up to 16 days): Eligibility for the study will be determined by Screening tests, physical examination/medical history, and fulfillment of eligibility criteria. Potential participants are required to provide written informed consent prior to the performance of any study specific Screening procedures.
* 2) Treatment Period (Day 1 to 57): Between 15 and 45 eligible male and female adult subjects will receive weekly RRx-001 for a total of nine doses and every other week nivolumab for a total of 5 doses (odd cycles) or 4 doses (even cycles). Study medication (RRx-001 and nivolumab) will be administered intravenously at the study center. The Treatment Period will end following the last dose of nivolumab. Subjects will attend the study center weekly for on-study assessments.
* 3) Follow-up Period: Subjects that have completed nivolumab dosing will undergo a follow-up assessment monthly, up to 100 days, for the emergence of delayed toxicity with particular attention to delayed immune related toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of an advanced, malignant, solid tumor(s) or lymphoma that are either refractory or is intolerant to, or has refused all standard available life-prolonging therapies.
* Measurable or evaluable disease based on RECIST criteria version. 1.1.
* ECOG performance status is 0-2 at Screening.
* Acceptable liver function at Screening,
* Serum creatinine < 2x institution upper limit of normal
* Acceptable hematologic status at Screening
* Female subjects of childbearing potential, and male subjects with partners of childbearing potential, must agree to use medically acceptable methods of contraception beginning on Study Day 1 and continuing until at least four weeks after administration of the subject's final dose of RRx-001.

Exclusion Criteria:

* Serious co-morbid medical condition, or a clinically significant laboratory finding(s) that, in the opinion of the Investigator, suggests the presence of an infectious, endocrine, and/or other inadequately treated systemic disorder.
* If female, subject is pregnant and/or breastfeeding.
* Subjects with active autoimmune disease or history of autoimmune disease that might recur and may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded.
* Subjects having a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.
* Prior therapy with any antibody/drug that targets the T cell coregulatory proteins, including but not limited to, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, and anti-CD40 antibodies. However, prior exposure to RRx-001 is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
Number, frequency and type of adverse events | 23 weeks

SECONDARY OUTCOMES:
Time to Tumor Progression (TTP) | 23 weeks
  Time to Tumor Progression (TTP) using Response Evaluation Criteria in Solid Tumors [RECIST v1.1] criteria
Overall Survival | 2 years
Clinical benefit Rate | 23 weeks
  Duration of clinical benefit (Stable disease or better) using Response Evaluation Criteria in Solid Tumors [RECIST v1.1] criteria
Progression-Free Survival (PFS) | 23 weeks
  Progression-Free Survival (PFS) using Response Evaluation Criteria in Solid Tumors [RECIST v1.1] criteria

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, MD, Study Director — EpicentRx, Inc.
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Reid T, Oronsky B, Caroen S, Quinn M, Williams J, Cabrales P, Abrouk N. Phase 1 pilot study of RRx-001 + nivolumab in patients with advanced metastatic cancer (PRIMETIME). Front Immunol. 2023 Mar 7;14:1104753. doi: 10.3389/fimmu.2023.1104753. eCollection 2023. PMID 36960054